CLINICAL TRIAL: NCT04068272
Title: Masked, Placebo Controlled, Phase I Trial to Assess the Safety of Bosentan 5 mg/ml Ophthalmic Eyewash in Type II Diabetic Patients
Brief Title: Safety of Bosentan in Type II Diabetic Patients
Acronym: BOSRET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Retinset SL (Industry)
Collaborators: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOBA-02-2016
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Bosentan

STUDY DESIGN:
Intervention Model Description: 1 Eye receives placebo, the other eye receives study drug. Eye elections is randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo and Study Drug have the same physical characteristics, labeling and packaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The patient will receive investigational product in one eye and placebo in the other eye. The allocation of treatment / placebo is masked and randomized
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator): The patient will receive investigational product in one eye and placebo in the other eye. The allocation of treatment / placebo is masked and randomized
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — Eyedrop
  Arms: Treatment
Drug: Placebo — Ophthalmic eyedrop with the exact same excipient of the drug arm without the active compound
  Arms: Placebo

SUMMARY:
This study evaluates the safety of topical Bosentan in Type II Diabetes patients

DETAILED DESCRIPTION:
The study is a Phase I, masked, placebo controlled clinical trial to assess safety of topical Bosentan in Type II Diabetes patients with no diabetes retinopathy

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Type II Diabetes Mellitus;
* 18 or more years old

Exclusion Criteria:

* Pregnant or breastfeeding Women
* Known allergy or intolerance to investigational product or any of its excipients
* Severe corneal abnormalities
* Any relevant ocular / ophthalmic pathology that may put study results at risk in the opinion of Principal Investigator
* Any sign or symptom of Diabetes Retinopathy
* Any ocular surgery in the 6 previous months to study inclusion
* Uncontrolled diabetes in the previous 3 months to inclusion or HbA1c levels ≥ 9% at baseline.
* Oxford Scale or OSDI scores compatible with study failure at inclusion visit. (Oxford ≥ 5 or OSTDI ≥ 13)
* Previous hepatopathy history or signs of hepatopathy at baseline.
* Contact lens use
* Actual treatment with the commercially available presentation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Epitheliopathy | 1 month
  Presence of epitheliopathy in the cornea or conjunctiva

SECONDARY OUTCOMES:
Presence of ocular discomfort | 1 month
  Presence of ocular discomfort assessed with Ocular Surface Disease Index (OSDI) questionnaire
Anterior segment inflammation | 1 month
  Presence of any sign of clinically significant inflammation at anterior segment

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - IOBA, Valladolid